CLINICAL TRIAL: NCT00643305
Title: HIV Prevention With the Mentally Ill: Motivation-Skills
Brief Title: HIV Prevention With the Mentally Ill
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Boston Medical Center (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Project HELP; 5R34MH075644-02 (NIH)
Record Dates: First submitted 2008-03-20; First posted 2008-03-26 (Estimated); Last update posted 2013-05-03 (Estimated); Status verified 2008-03

CONDITIONS: HIV Infections
Keywords: HIV; Motivational Interviewing; Skills; Prevention; Mental illness; Risk reduction; HIV/AIDS; HIV Seronegativity
MeSH Terms: conditions — HIV Infections; Mental Disorders; Risk Reduction Behavior; Acquired Immunodeficiency Syndrome | interventions — Motivational Interviewing

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Skills Building with Motivational Interviewing (SB-MI)- combines education and general skills-building participants can use to reduce their at-risk behavior for HIV with increasing motivation to change HIV risk behaviors
  Interventions: Behavioral: Skills Building with Motivational Interviewing
- 2 (Active Comparator): Skills Building (SB) - provides education and general skills-building for reduction of HIV risk behaviors.
  Interventions: Behavioral: Skills Building

INTERVENTIONS:
Behavioral: Skills Building with Motivational Interviewing — Based on the Stages of Change model, participants are provided with feedback related to their current HIV risk and Motivational Interviewing strategies are used to increase motivation to decrease HIV risk behaviors. Participants are also provided with information and training in skills critical for reducing HIV risk
  Arms: 1
Behavioral: Skills Building — Participants are provided with information and training in skills critical for reducing HIV risk.
  Arms: 2

SUMMARY:
The purpose of this study is to determine whether motivational interviewing and skills building interventions reduce HIV risk behavior for adults with serious and persistent mental illness.

DETAILED DESCRIPTION:
Our long-term objective is to reduce the incidence of HIV for people with serious and persistent mental illness (SMI) by developing an effective primary and secondary HIV risk reduction intervention for this population which can be easily delivered in the "real world" settings in which patients routinely receive care. Research findings document that the incidence of HIV infection, sexually transmitted diseases, and sexual and drug use behaviors are high among people with serious mental illness, as evidenced by rates of HIV infection and other sexually-transmitted diseases (STDs). A variety of factors underlie risky behaviors for the SMI, including cognitive impairment, poor judgment, affective instability and impulsiveness.

Skills-building (SB) HIV risk reduction interventions, typically delivered in a small group formats, have had modest success in increasing HIV-related knowledge and improving risk reduction skills for people with SMI, although these effects are transient. As skills-building interventions are currently the standard of care in most research and clinical settings for HIV prevention, it is important to identify new ways to augment these interventions.

A relatively new and promising addition to the armamentarium of individualized interventions is Motivational Interviewing (MI). MI is an approach designed to reduce ambivalence and enhance intrinsic motivation to change problematic behaviors. Previous researchers have noted effects for both SB and MI interventions independently, however, these effects tend to be fairly modest. Integrating these approaches in a systematized way allows us to test the degree to which this combination is useful, given that both motivation and skills are clearly important in effecting health behavior change.

Our specific primary aims are the following:

1. To adapt SB and MI interventions for HIV risk reduction for men and women with serious and persistent mental illness (SMI).

   Interventions for HIV risk reduction for people with SMI are typically offered in a group format and focus primarily on skills-building. We have developed and refined a brief, individually-tailored skills-building intervention (SB Intervention), based on these existing manuals. We have also adapted and refined a brief individually-tailored Motivational Interviewing intervention to target HIV risk behaviors, incorporating skills-building techniques analogous to those in the SB intervention, resulting in a Motivational-Interviewing & Skills-Building Intervention (SB-MI Intervention). Adaptation and refinement of the SB and SB-MI interventions was informed by consulting with experts in MI, SMI, and HIV risk reduction, eliciting feedback from advisory boards of providers and consumers, and conducting feedback interviews with participants who have completed participation in the study.
2. To pilot test and obtain preliminary data with regard to the feasibility of our interventions and the differences in outcome associated with our SB and SB-MI interventions for reduction of HIV-related risk behaviors in a cohort of SMI adults.

   Comparison of SB and SB-MI interventions in the proposed pilot study will allow us to assess the degree to which incorporation of motivational techniques are helpful in augmenting skills-building interventions for HIV risk reduction for people with SMI. These preliminary analyses will inform our need to refine the adapted interventions (SB and SB-MI).
3. To offer HIV counseling and testing for at-risk individuals with SMI, with an emphasis on connecting participants to appropriate medical and mental health services.

   To date, increasing rates of HIV counseling and testing for the SMI has not been a primary focus of clinical research, which we believe to be a significant public health deficit. As part of both of our interventions we are providing information about HIV counseling and testing services to those participants not identified as HIV-seropositive and encouraging them to access these services. We are then tracking the degree to which participants follow up on these referrals as part of our follow-up evaluations. This will allow us to test the degree to which our interventions are helpful in increasing rates of HIV testing.
4. To begin to explore the relationships between participant characteristics, HIV risk behaviors, and response to our interventions.

One of the unique features of our intervention is that it assumes an individually-tailored approach, which can address unique patient characteristics inherent in a heterogeneous sample. Indeed, using a heterogeneous sample greatly facilitates our primary long-term objective, which is to develop useable interventions that can be adapted in real-world settings. This project will allow us to begin to identify those characteristics that are likely to be associated with more positive outcomes (i.e. greater risk reduction, increased rates of HIV testing).

ELIGIBILITY:
Inclusion Criteria:

* Age 19 and older
* Able to provide consent
* Able to understand and speak English
* Willing and able to participate
* Suffer from a serious and persistent mental illness (SMI)
* Have had at least one HIV risk behavior (unprotected sexual activity, sharing injection drug needles without following Center for Disease Control guidelines for needle-cleaning, sexual activity while under the influence of drugs or alcohol) during the three-month period prior to the baseline evaluation

Exclusion Criteria:

* Do not suffer from a serious mental illness
* Have not engaged in an HIV risk behavior during the three-month period prior to the baseline evaluation.
* Unable to provide consent
* Unable to understand and speak English
* Under the age of 19

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2006-02; Primary Completion 2008-10 (Actual); Study Completion 2009-01 (Actual)

PRIMARY OUTCOMES:
Self-reported reduction in HIV risk behavior for infection/re-infection of HIV, as measured by administration of the TimeLine Follow-Back. | 6 months
Skillfulness in behaviors critical for efficacious use of HIV risk reduction strategies, measured by standardized role-plays and demonstrations | 6 months
HIV-related knowledge, as measured by the HIV Knowledge Questionnaire (HIV-KQ) | 6 months
Accessing HIV counseling and testing, assessed by self-report | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Brady, Ph.D., Principal Investigator — The Trustees of Boston University, BUMS
Locations (1):
- Boston Medical Center, Boston, Massachusetts, United States